CLINICAL TRIAL: NCT02714920
Title: DNA Repair Enzyme Signature Associated With Response to Chemo- and Radio-therapy in Head and Neck Cancer: ChemRadAssay
Brief Title: DNA Repair Enzyme Signature in Head and Neck Cancer (CHEMRAD)
Acronym: CHEMRAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL15_0188; 2015-A00911-48 (Other: ANSM)
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Head Cancer; Neck Cancer
Keywords: DNA Repair Enzyme Signature; instrinsic radio- or chemo-resistance; treatment-induced radio- or chemo-resistance
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DNA Repair enzyme signature (Other): Tumor biopsies and blood samples performed specifically to determine DNA Repair enzyme signature biomarkers profiles (CHEMRAD assay)
  Interventions: Other: CHEMRAD assay

INTERVENTIONS:
Other: CHEMRAD assay — CHEMRAD is a new biomarker research strategy based on three assays that enables the functional characterization of DNA repair capacities.

SUMMARY:
Squamous cell carcinoma (HNSCC) is the most frequent form of head and neck cancer. The therapeutic choice depends on the stage of the disease and the habits of the medical teams. Surgery, radiotherapy and chemotherapy can be used, alone or combined. However, none of the existing strategies has proven its superiority.

Chemotherapy and radiotherapy induce DNA damages in the tumor cells. However, cells have the ability to induce DNA reparation, capable of causing treatment resistance. DNA reparation in non-tumor tissues can also explain the toxicity of cancer treatments.

Investigation of DNA repair pathways involved in chemo- or radiation resistance could offer a good strategy for identifying biomarkers or indicators of treatment response. This study will explore the capacity of a comprehensive functional approach that addresses several pathways, based on the use of three innovative patented technologies, to classify the tumor response of HNSCC patients to treatments according to their DNA Repair Enzyme Signature.

Our hypothesis is that taking into account various clinical parameters (e.g. patient and tumor characteristics), treatment strategy and measuring the DNA Repair Enzyme Signature would create patients' profiles and optimize their management.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old;
* HNSCC proven on a biopsy, located in the oral cavity or the oropharynx (the tumor must be accessible to a biopsy during an outpatient visit);
* Tumor accessible to a biopsy under local anesthesia;
* TNM classification: any stage except M1;
* Eligible for radiotherapy as a curative treatment;
* No surgery planned as exclusive treatment;
* Able to comply with the scheduled visits;
* Affiliated to or beneficiary of a social security system (or equivalent) ;
* Having given written informed consent prior to any procedure related to the study.

Exclusion Criteria:

* Recurrence or second cancer in a previously irradiated area;
* Nasopharyngeal carcinoma;
* Tumor requiring general anesthesia to perform the biopsy;
* Radiotherapy planned to be provided outside of the investigation center;
* Pregnant or lactating woman;
* Adult ward of court (under guardianship or trusteeship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
DNA Repair Enzyme Signature biomarkers profiles according to intrinsic or treatment-induced radio- or chemo-resistance in different tumor and clinical settings. | 18 months after the end of the treatments (approximately 24 months after the beginning of the study)
  Results of DNA Repair Enzyme biomarker profiles of tumor cells will be quantified before and during treatment with:
  * The excision/synthesis assay, as the incorporated fluorescence intensity;
  * The ODN (Oligonucleotide) assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB (Double-strand breaks) Assay, as the incorporated fluorescence intensity.
  The radio- or chemo-resistance will be defined as disease-free survival, i.e. absence of local or regional recurrence in irradiated tissue seen on CT-scan.
  The different tumor and clinical settings will be determined with:
  * Patient and tumor characteristics, i.e. age, sex, etiological factors (tobacco, alcohol), localization and stage of the tumor, HPV (Human Papilloma Virus) status, p53 status;
  * Treatment strategy, i.e. all the treatments that will be administered to the patient and their sequence, including International Nonproprietary Name of the drugs and doses of chemo and/or radiotherapy

SECONDARY OUTCOMES:
DNA Repair Enzyme Signature biomarkers profiles according to instrinsic or treatment-induced radio- or chemo-resistance. | 4 months after the end of the treatments (approximately 10 months after the beginning of the study)
  Results of DNA Repair Enzyme biomarker profiles of tumor cells will be quantified before and during treatment with:
  * The excision/synthesis assay, as the incorporated fluorescence intensity;
  * The ODN assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB Assay, as the incorporated fluorescence intensity. The radio- or chemo-resistance will be defined as disease-free survival, i.e. absence of local or regional recurrence in irradiated tissue measured on the CT-scan performed 4 months after the end of the treatment.
DNA Repair Enzyme Signature biomarkers profiles according to tumor response to treatment | 4 months after the end of the treatments (approximately 10 months after the beginning of the study)
  Results of DNA Repair Enzyme biomarker profiles of tumor cells will be quantified before and during treatment with:
  * The excision/synthesis assay, as the incorporated fluorescence intensity;
  * The ODN assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB Assay, as the incorporated fluorescence intensity. Global response to treatment measured on the CT-scan according to RECIST criteria, at 4 months after the end of the treatment.
DNA Repair Enzyme Signature biomarkers profiles according to tumor response to treatment | 18 months after the end of the treatments (approximately 24 months after the beginning of the study)
  Results of DNA Repair Enzyme biomarker profiles of tumor cells will be quantified before and during treatment with:
  * The excision/synthesis assay, as the incorporated fluorescence intensity;
  * The ODN assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB Assay, as the incorporated fluorescence intensity. Global response to treatment measured on the CT-scan according to RECIST criteria, at 18 months, after the end of the treatment.
DNA Repair Enzyme Signature biomarkers profiles according to immediate treatment-induced toxicity | At the end of the treatments (an average of 6 months after the beginning of the study)
  Results of DNA Repair Enzyme biomarker profiles of tumor cells will be quantified before and during treatment with:
  * The excision/synthesis assay, as the incorporated fluorescence intensity;
  * The ODN assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB Assay, as the incorporated fluorescence intensity. Treatment-induced adverse events occurring during the treatment.
DNA Repair Enzyme Signature biomarkers profiles of Peripheral Blood Mononuclear Cells (PBMCs). | 4 months after the end of the treatment (approximately 10 months after the beginning of the study)
  Results of DNA repair enzyme signature of Peripheral Blood Mononuclear Cells quantified before and during treatment with:
  * The ODN assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB Assay, as the incorporated fluorescence intensity.
DNA Repair Enzyme Signature biomarkers profiles of Peripheral Blood Mononuclear Cells (PBMCs). | 18 months after the end of the treatment (approximately 24 months after the beginning of the study)
  Results of DNA repair enzyme signature of Peripheral Blood Mononuclear Cells quantified before and during treatment with:
  * The ODN assay, as the percentage of cleavage for the DNA target lesions;
  * The DSB Assay, as the incorporated fluorescence intensity.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Grenoble - Hôpital Michallon, Grenoble
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Pierre-Bénite